CLINICAL TRIAL: NCT03404050
Title: A Community Based Music and Dance Movement Therapy Group for Older Adults With Dementia
Brief Title: Community Based Music and Dance Movement Therapy Group for Older Adults With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edge Hill University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL PhD
Record Dates: First submitted 2018-01-09; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Assessments taken at three different time periods: week zero, week five and week eleven.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music and dance movement therapy group (Experimental): Music and dance movement therapy group
  Interventions: Other: Music and dance movement therapy

INTERVENTIONS:
Other: Music and dance movement therapy — Theoretically, the intervention adopts a humanistic approach of person centred care highlighting the importance of maintaining and enhancing personhood for older people with dementia.

SUMMARY:
This study explores the value of a particular community based music and dance movement therapy group for older adults with dementia?

To answer this question, the investigators intend to address the following two sub-questions:

1. How does participants' use of music and movement change over time?
2. Did a music and dance movement therapy group improve participants' depressive symptoms?

DETAILED DESCRIPTION:
A systematic review identified a need to explore the value of an arts therapies group for older adults with dementia living in the community with early to moderate stage dementia. This client population commonly experience depression, social withdrawal and cognitive difficulties and literature suggests a music and dance movement therapy group could potentially make a contribution to both reducing symptoms and improving communication and wellbeing. However, there is still lack of clarity on clinically meaningful outcome measures, detail regarding the therapeutic process and questions remain regarding the trustworthiness of qualitative observations. This mixed method feasibility study aims to test whether the interventions translate to a community setting, provide richer insight into the meaningful aspect of the therapeutic process and provide some preliminary quantitative findings.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old
* Living in the community
* Diagnosis of dementia
* Adequate functional hearing/vision
* Sufficient knowledge of English to understand participant information sheet

Exclusion Criteria:

* Participants excluded if they suffered from any physical or psychological conditions that make it difficult to access a group setting independently.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Cornell Scale for Depression in Dementia | 7 days
  Joint interview with participant and care provider/family member regarding signs and symptoms of depression; a score greater than 10 indicates probably major depressive episode

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Karkou, Study Director — Edge Hill University
Locations (1):
- Edge Hill University, Ormskirk, Lancs, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Registered systematic review protocol — http://www.crd.york.ac.uk/PROSPERO/display_record.asp?ID=CRD42015029463